CLINICAL TRIAL: NCT02367196
Title: A Phase I, Open-Label, Dose Finding Study of CC-90002, a Monoclonal Antibody Directed Against CD47, in Subjects With Advanced Solid and Hematologic Cancers
Brief Title: A Phase 1, Dose Finding Study of CC-90002 in Subjects With Advanced Solid and Hematologic Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-90002-ST-001; 2015-000101-39 (EudraCT Number)
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Hematologic Neoplasms
Keywords: CC-90002; Monoclonal; Antibody; CD47; Advanced; Solid Cancers; Hematologic Cancers
MeSH Terms: conditions — Hematologic Neoplasms | interventions — CC-90002; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A: CC-90002 (Experimental): CC-90002 will be given by intravenous (IV) infusion on a 28 day cycle
  Interventions: Drug: CC-90002
- Part B: CC-90002 with Rituximab (Experimental): CC-90002 in combination with Rituximab will be given by intravenous (IV) infusion on a 28 day cycle in subjects with CD20-positive NHL
  Interventions: Drug: CC-90002; Drug: Rituximab

INTERVENTIONS:
Drug: CC-90002
Drug: Rituximab
  Arms: Part B: CC-90002 with Rituximab

SUMMARY:
CC-90002-ST -001 is an open-label, Phase 1, dose escalation clinical study in subjects with advanced, refractory solid and hematologic cancers.

DETAILED DESCRIPTION:
CC-90002-ST-001 is an open-label, Phase 1, dose escalation, first in human (FIH) clinical study of CC-90002, administered by intravenous (IV) infusion, in subjects with advanced, refractory solid and hematologic cancers.

The study will be conducted in two parts. Part A dose escalation phase will explore escalating dose cohorts of the study drug CC-90002.

Part B dose escalation will explore escalating doses of CC-90002 in combination with rituximab in subjects with CD20-positive NHL.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, 18 years or older, with advanced, relapsed or refractory solid tumors, Multiple Myeloma (MM) or non-Hodgkin's lymphoma (NHL) in Part A. In Part B, relapsed and/or refractory CD20-positive NHL subjects only.
2. At least one site of measurable disease in subjects with solid tumors and NHL.
3. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
4. Subjects must have adequate hematopoietic, liver, renal and coagulation function as assessed by specific laboratory criteria.
5. Females and males must agree to contraceptive methods and avoid conceiving throughout the study, and for up to 8 weeks following the last dose of CC-90002. If participating in Part B, females of child bearing potential should continue to use effective contraceptive methods for 12 months following treatment with rituximab

Exclusion Criteria:

1. High grade lymphomas (Burkitts or lymphoblastic), plasma cell leukemia.
2. High grade, rapidly proliferative solid tumors (eg, small cell lung cancer, germ cell tumors, neuroblastoma) with extensive tumor burden.
3. Symptomatic central nervous system involvement.
4. Impaired cardiac function or clinically significant cardiac disease.
5. Prior Red blood cell (RBC) transfusion < 3 months prior to starting CC-90002 (Part A only).
6. Prior autologous stem cell transplant ≤ 3 months prior to starting CC-90002.
7. Prior allogeneic stem cell transplant with either standard or reduced intensity conditioning ≤ 6 months prior to starting CC-90002.
8. Prior systemic cancer-directed treatments or investigational modalities ≤ 5 half lives or 4 weeks prior to starting CC-90002, whichever is shorter.
9. Major surgery ≤ 2 weeks prior to starting CC-90002.
10. Pregnant or nursing females.
11. Known HIV infection.
12. Known chronic, active hepatitis B or C (HBV/HCV) infection.
13. Ongoing treatment with chronic, therapeutic dosing of anti-coagulants.
14. History of autoimmune hemolytic anemia or autoimmune thrombocytopenia.
15. History of concurrent second cancers requiring active, ongoing systemic treatment.

concurrent second cancers requiring active, ongoing systemic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03-12 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | Up to 18 months
  Number of participants with a DLT
Non-Tolerated Dose (NTD) - Part A | Up to 18 months
  Dose at which 2 or more of up to 6 evaluable subjects in any dose cohort experience a DLT in Cycle 1.
Maximum Tolerated Dose (MTD) - Part A | Up to 18 months
  Dose that is the last dose level below the NTD with 0 or 1 out of 6 evaluable subjects experiencing a DLT during Cycle 1.
Non-Tolerated Dose (NTD) - Part B | Up to 24 months
  Dose at which 2 or more of up to 6 evaluable subjects in any dose cohort experience a DLT in Cycle 1.
Maximum Tolerated Dose (MTD) - Part B | Up to 24 months
  Dose that is the last dose level below the NTD with 0 or 1 out of 6 evaluable subjects experiencing a DLT during Cycle 1.

SECONDARY OUTCOMES:
Antitumor efficacy | Up to 36 months
  Determined by response rates of each tumor type using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and other tumor-appropriate response criteria.
Pharmacokinetics - Cmax | Cycle 1 and beyond; and after discontinuation
  Maximum observed concentration in serum
Pharmacokinetics - AUC | Cycle 1 and beyond; and after discontinuation
  Area under the serum concentration - time curve
Pharmacokinetics - tmax | Cycle 1 and beyond; and after discontinuation
  Time to peak (maximum) serum concentration
Pharmacokinetics - T1/2 | Cycle 1 and beyond; and after discontinuation
  Terminal half-life (T1/2)
Pharmacokinetics - CL | Cycle 1 and beyond; and after discontinuation
  Total body clearance of the drug from serum
Pharmacokinetics - Vmax | Cycle 1 and beyond; and after discontinuation
  Volume of distribution at steady-state
Anti-Drug Antibodies (ADAs) | Cycle 1 and beyond; and after discontinuation
  Determine the presence and frequency of anti-drug antibodies
Overall Survival - Part B | Up to 2 years
  Measured as the time from the first dose of CC-90002 to death due to any cause.
Progression-free survival- Part B | Up to 2 years
  Defined as the time from the first dose of CC-90002 to the first occurrence of disease progression or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Michael Burgess, MD, PhD, Study Director — Celgene
Locations (13):
- United States (5):
  - Scottsdale Healthcare Research Institute, Scottsdale, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - University of California San Francisco, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
- Spain (8):
  - Hospital Universitari Germans Trias i Pujol Can Ruti, Badalona (Barcelona)
  - Hospital Val d'Hebron, Barcelona
  - Duran i Reynals Institut Catala d'Oncologia, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Marques de Valdecilla, Santander
  - Hospital de la Fe, Valencia

REFERENCES:
- [Derived] Narla RK, Modi H, Bauer D, Abbasian M, Leisten J, Piccotti JR, Kopytek S, Eckelman BP, Deveraux Q, Timmer J, Zhu D, Wong L, Escoubet L, Raymon HK, Hariharan K. Modulation of CD47-SIRPalpha innate immune checkpoint axis with Fc-function detuned anti-CD47 therapeutic antibody. Cancer Immunol Immunother. 2022 Feb;71(2):473-489. doi: 10.1007/s00262-021-03010-6. Epub 2021 Jul 10. PMID 34247273